CLINICAL TRIAL: NCT00548067
Title: A Multi-center, Multiple Dose, Open-label, Four-cohort, Parallel Study to Assess the Pharmacokinetic Drug Interaction Following Co-administration of Valsartan, Hydrochlorothiazide and Amlodipine in Patients With Hypertension.
Brief Title: Pharmacokinetic Drug Interaction Study Following Co-administration of Valsartan, Hydrochlorothiazide and Amlodipine in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVEA489A2104
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Hypertension
Keywords: High blood pressure, hypertension, drug interaction, steady state, valsartan, hydrochlorothiazide, amlodipine
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide; Amlodipine, Valsartan Drug Combination; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: Valsartan/hydrochlorothiazide (HCTZ)
- 2 (Active Comparator)
  Interventions: Drug: Valsartan/amlodipine
- 3 (Active Comparator)
  Interventions: Drug: Amlodipine/hydrochlorothiazide(HCTZ)
- 4 (Experimental)
  Interventions: Drug: Valsartan/amlodipine/hydrochlorothiazide(HCTZ)

INTERVENTIONS:
Drug: Valsartan/hydrochlorothiazide (HCTZ)
  Arms: 1
Drug: Valsartan/amlodipine
  Arms: 2
Drug: Amlodipine/hydrochlorothiazide(HCTZ)
  Arms: 3
Drug: Valsartan/amlodipine/hydrochlorothiazide(HCTZ)
  Arms: 4

SUMMARY:
The purpose of this study is to determine potential pharmacokinetic drug-drug interaction when three drugs (valsartan, amlodipine, and hydrochlorothiazide) are co-administered.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed as hypertensive

* Untreated confirmed hypertensive patients (consistent SBP >140 mm Hg or DBP >90 mm Hg)
* Uncontrolled hypertensive patients (Consistent SBP >140 mm Hg or DBP >90 mm Hg) on one drug therapy.
* Uncontrolled hypertensive patients (Consistent SBP >140 mm Hg or DBP >90 mm Hg) on two drug therapy.

Exclusion Criteria:

* Inability to switch from all prior antihypertensive medications safely as required by the protocol.
* Need for drugs other than study drugs at the time of baseline.
* Patients with SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg at screening.
* Patients on four or more antihypertensive drugs at screening.
* Pregnant or nursing (lactating) women.
* Patients with diabetes mellitus
* Patients with heart diseases and any other disease

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2007-09; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Potential drug interaction and effect on blood level of drugs when co-administered for 17 days

SECONDARY OUTCOMES:
Safety and tolerability of co-administered assessed by capturing adverse events and safety laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigative site
Locations (5):
- India (5):
  - Novartis Investigative Site, Ahmedabad
  - Novartis investigative site, Bangalore
  - Novartis Investigative site, Hyderabad
  - Novartis Investigative site, Mangalore
  - Novartis investigative site, Mehasana